CLINICAL TRIAL: NCT07213154
Title: Assessment of Novel Label-free Optical Imaging Technology for the Evaluation of Skin Lesions
Brief Title: Optical Imaging Scans for the Diagnosis of Skin Cancer in Patients With Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mohammad K. Khan, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00008502; NCI-2025-02356 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00008502 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6407-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2025-08-26; First posted 2025-10-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Malignant Skin Neoplasm; Skin Disorder; Skin Neoplasm
MeSH Terms: conditions — Skin Neoplasms; Skin Diseases | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group I (qOBM) (Experimental): Patients who have skin melanoma and/or suspected dysplastic nevi undergo qOBM optical imaging scan on study. Patients may undergo 2 additional qOBM optical imaging scans at the discretion of the treating physician. After qOBM scans, patients who are diagnosed with skin cancer may proceed to Group II.
  Interventions: Procedure: Quantitative Oblique Back-Illumination Microscopy
- Group II (qOBM, SOC RT) (Experimental): GROUP II: Patients with skin cancer who are undergoing SOC RT undergo qOBM optical imaging scans prior to- and during or after SOC RT on study. Patients may also undergo qOBM optical imaging scans additional at approximately 1, 6, and 12 months after completion of SOC RT at the discretion of the treating physician.
  Interventions: Procedure: Quantitative Oblique Back-Illumination Microscopy; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Quantitative Oblique Back-Illumination Microscopy — Undergo qOBM
  Other Names: qOBM
Radiation: Radiation Therapy — Undergo SOC RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Group II (qOBM, SOC RT)

SUMMARY:
This clinical trial studies how well an optical imaging scan called quantitative oblique back-illumination microscopy (qOBM) helps in diagnosing skin cancer in patients with skin lesions. qOBM is a non-invasive procedure that uses red light for illumination, and may work better than no imaging procedures in aiding doctors in diagnosing skin lesions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To perform a first-in-human study to assess the ability of a qOBM handheld device to reliably image skin pathology in-situ and in-vivo.

SECONDARY OBJECTIVES:

I. Characterize a wide variety of lesions including but limited to:

Ia. Malignant lesions: basal cell cancers, squamous cell cancers, Merkel cell cancer, melanoma, etc,; Ib. Non-malignant lesions: keloids, surgical scars, actinic keratosis, benign and dysplastic nevi, cysts, lipoma; Ic. Inflammatory conditions: psoriasis, eczema, alopecia, acne, wounds, etc); Id. Characterize pre and post treatment changes in the lesion as well as the surrounding normal tissue stroma (examples, but not limited to: changes to hair follicles, epidermis, dermis, subcutaneous tissue, erector pillae muscles, vessels, nerves, etc); Ie. Correlate optical findings with histological findings for lesions that would have been removed surgically and/or are biopsied (examples, but not limited to: removal of a skin cancer where optical imaging is used to characterize peripheral extent of the lesion as well as depth of penetration, a benign versus malignant lesion, pigmented versus [vs] non-pigmented lesion, etc).

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients who have skin melanoma and/or suspected dysplastic nevi undergo qOBM optical imaging scan on study. Patients may undergo 2 additional qOBM optical imaging scans at the discretion of the treating physician. After qOBM scans, patients who are diagnosed with skin cancer may proceed to Group II.

GROUP II: Patients with skin cancer who are undergoing standard of care (SOC) radiation therapy (RT) undergo qOBM optical imaging scans prior to- and during or after SOC RT on study. Patients may also undergo qOBM optical imaging scans additional at approximately 1, 6, and 12 months after completion of SOC RT at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Candidate with skin lesions
* Signed study-specific informed consent prior to study entry
* ≥ 18 years old

Exclusion Criteria:

* Prior surgery or radiotherapy to the area to be treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2027-09-17 (Estimated)

PRIMARY OUTCOMES:
qOBM Clinical Assessment | Up to 12 months
  Assessing the application of quantitative oblique back-illumination microscopy (qOBM) to assess skin pathology. Analysis will be descriptive in nature (e.g., appearance of cells in the epidermis, dermis, and basal junction). Quantitative analysis will include extracting image features such as mean, standard deviation, and kurtosis of the phase values; entropy, fractal dimension, gray level co-occurrence matrix, and other mathematical image features. Radiation Therapy Oncology Group (RTOG) Acute Radiation Morbidity Scoring Criteria (Skin) Grade 0. No change over baseline, Grade 1. Follicular, faint or dull erythema/epilation/dry desquamation/decreased sweating, Grade 2. Tender or bright erythema, patchy moist desquamation/moderate edema, Grade 3. Confluent, moist desquamation other than skin folds, pitting edema, Grade 4. Ulceration, hemorrhage, necrosis

SECONDARY OUTCOMES:
Usability of the qOBM Device | Up to 12 months
  Will collect information regarding the usability of the device, including how ergonomic it is, ideal for factors for acquiring images and visualizing structures in real time. Quantitative analysis will include extracting image features such as mean, standard deviation, and kurtosis of the phase values; entropy, fractal dimension, gray level co-occurrence matrix, and other mathematical image features. Differences between similar diagnoses vs adjacent normal skin will be evaluated using a two-sided t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad K. Khan, MD, PhD, MS, FACRO, FACR, DABR, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia